CLINICAL TRIAL: NCT00229307
Title: Prolonged Exposure (PE) Treatment for Post Traumatic Stress Disorder (PTSD) 20 Minutes Versus 40 Minutes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-05-3709-JZ-CTIL
Record Dates: First submitted 2005-09-28; First posted 2005-09-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: PTSD
Keywords: Post traumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Behavioral: Prolonged Exposure (PE) therapy
- 2 (Active Comparator)
  Interventions: Behavioral: Prolonged Exposure (PE) therapy

INTERVENTIONS:
Behavioral: Prolonged Exposure (PE) therapy — 20 minutes exposure
  Arms: 1
Behavioral: Prolonged Exposure (PE) therapy — 40 minutes exposure
  Arms: 2

SUMMARY:
Comparing the efficacy of 40 minutes PE treatment to 20 minutes of the same treatment

ELIGIBILITY:
Inclusion Criteria:

* PTSD

Exclusion Criteria:

* Psychotic symptoms
* Dissociation
* Drug or Alcohol dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
PSS-i | 15 weeks and 1-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nitza Nacasch, MD, Study Chair — Sheba Medical Center; Joseph Zohar, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel